CLINICAL TRIAL: NCT02761811
Title: A Prospective, Multicenter, Single Blind, Randomized and Sham Controlled Trial of Renal Sympathetic Denervation Using SyMapCath I™ Catheter and SYMPIONEER S1™ Stimulator/Generator for the Treatment of Hypertension (SMART Trial)
Brief Title: Sympathetic Mapping/ Ablation of Renal Nerves Trial
Acronym: SMART
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SyMap Medical (Suzhou), Ltd. (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-01
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Radionuclide Generators

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal Sympathetic Denervation (Experimental): Percutaneous renal denervation using the SyMapCath I™ Catheter and SYMPIONEER S1™ Stimulator/Generator.
  Interventions: Device: SyMapCath I™ catheter and SYMPIONEER S1™ Stimulator/Generator
- Masked Procedure (Sham Comparator): Percutaneous renal artery angiography
  Interventions: Device: SyMapCath I™ catheter and SYMPIONEER S1™ Stimulator/Generator

INTERVENTIONS:
Device: SyMapCath I™ catheter and SYMPIONEER S1™ Stimulator/Generator — Radiofrequency ablation of renal arterial sympathetic nerves

SUMMARY:
To evaluate the safety and efficacy of targeted renal sympathetic denervation using SyMapCath I® and SYMPIONEER S1® Stimulator/ Generator in patients with essential hypertension for at least 6 months of the disease history and pharmacotherapy, however, their blood pressure still cannot be controlled, then after standardized antihypertensive drug therapy (at least two drugs) for at least 28 days, office systolic blood pressure is still ≥ 150mmHg, ≤180mmHg.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single blind, randomized and sham controlled trial, in which patients are diagnosed with essential hypertension with at least six months of the disease history and pharmacotherapy however their blood pressure still cannot be controlled. The patients will be informed, consent and get into a screening process. During the screening period patients will receive a standardized antihypertensive drug treatment for at least 28 days and office systolic blood pressure is still ≥ 150mmHg, ≤180mmHg, and meet the inclusion and exclusion criteria. These patients will conduct renal artery angiography and be allocated to either renal sympathetic nerve denervation group or renal artery angiography group by a randomizing system in a 1:1 ratio (220 patients, 110 pairs). Patients with office systolic blood pressure which is not achieved ideal level (<140 mmHg) will titrate doses or classes of antihypertensive drugs according to a predefined standardized medication regimen until their office systolic blood pressure <140 mmHg, whereas in principle patients should follow the drug titration regimen, however, it is allowed to adjust antihypertensive medications per the real-world needs after 12 months.

Physicians who perform post-procedure patient management and physicians who perform renal denervation procedures are blinded to each other.

Patients will be followed at 7 days after the procedure or at discharge from hospital, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 9 months, 12months, 24months, 36 months, 48 months and 60 months for blood pressure measurements and antihypertensive medications. Urine samples will be collected for drug tests (LC-MS/MS) to determine drug compliance of a patient by an independent laboratory.

Data collecting/management/statistical analysis and laboratory tests will be done by independent, qualified organizations. Independent DSMB/CEC are formed and responsible for assessments of protocol deviations and natures of SAEs.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant female subjects, 18≤age≤65
2. Essential hypertension
3. Office systolic blood pressure ≥150mmHg and ≤180mmHg; and resting heart rate ≥70 bpm without taking beta blocker(Resting heart rate does not taken into account if beta blocker is taken)
4. Average 24-hour ABPM systolic blood pressure ≥130mmHg, or ABPM systolic blood pressure during daytime ≥ 135mmHg, or ABPM systolic blood pressure during nighttime ≥ 120mmHg
5. History of hypertension is longer than 6 months
6. Patient with poor blood pressure control after 6 months of antihypertensive drug therapy, understands the purpose of this study, and is willing to participate and sign the Informed Consent; then the patient receives standard antihypertensive drug treatment (at least two drugs) for at least 28 days, drug compliance ≥80%, office systolic blood pressure ≥150 mmHg and ≤180 mmHg.
7. Patient is compliant and willing to complete clinical follow-up.

Exclusion Criteria:

1. Renal artery anatomy is unqualified including： (1) diameter <4mm or treatable length <25mm， (2) multiple renal arteries and the main renal artery supplies a fraction of the blood flow less than 75%, (3) renal artery stenosis >50% or any renal artery aneurysms on either side, (4) history of renal artery PTA, including balloon angioplasty and stenting.
2. eGFR <45mL/min/1.73m2 (MDRD formula)
3. Hospitalized within one year due to hypertensive crisis
4. Average 24-hour systolic blood pressure <130mmHg and ABPM systolic blood pressure during daytime ≤ 135mmHg, and ABMP systolic blood pressure during nighttime ≤ 120mmHg
5. Pulse pressure >80mmHg
6. During running in period, using antihypertensive drugs other than standardized antihypertensive drugs
7. Participated other clinical trials including both drug and medical device studies within 3 months from current study
8. Female with pregnant or lactating, or having plans for pregnancy within 1 year
9. Patient with sleep apnea who needs chronic oxygen-breathing or mechanical ventilation support (for example, tracheostomy)
10. Patients previously or currently suffering from following diseases:

(1) essential pulmonary arterial hypertension, (2) type I diabetes, (3) patients with severe cardiac valvular stenosis who have contradictions and cannot rolerant to significantly reduce blood pressure, (4) within half year, patients had myocardial infraction, unstable angina, syncope or cerebrovascular accidents, (5) history of primary aldosteronism, pheochromocytoma, aorta stenosis, hyperthyroidism or hyperparathyreosis, (6) any disease conditions interfering the measurement of blood pressure (for instance, severe peripheral artery diseases, abdominal artery aneurysm, hemorrhagic disorders such as thrombocytopenia, hemophilia and severe anemia), (7) plans to have surgery or cardiovascular interventions within 6 months, (8) alcohol abuse or unknown drug dependence history, (9) neuroticisms such as depression or anxiety disorders, (10) non-compliant patients who are unable to follow the study protocol per physician's requests.

11. Any contradictions to conduct renal artery stimulation and ablation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-06-30; Primary Completion 2022-08-25 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The control rate of office systolic blood pressure ( SBP<140mmHg) | 6 months after the treatment
  The control rate of office systolic blood pressure ( SBP<140mmHg) at 6 months after the treatment
Change in the composite index of antihypertensive drugs to reach control of office systolic blood pressure (<140mmHg) | 6 months after the treatments
  Change in the composite index of antihypertensive drugs to reach control of office systolic blood pressure (<140mmHg) at 6 months after the treatment

SECONDARY OUTCOMES:
Reduction in average 24-hour Ambulatory Blood Pressure Monitoring (ABPM) systolic blood pressure | 6 months
Postoperative reduction in 24-hour ABPM in systolic, diastolic and mean arterial blood pressure | discharge day or 7 days after procedure
Reduction in office blood pressure | 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 12 months, 24months, 36 months, 48 months and 60 months
Change in composite index of antihypertensive drugs | 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, 12 months, 24months, 36 months, 48 months and 60 months
Success rate of the renal interventional therapy procedure | during the procedure
  the renal denervation catheter can be engaged to the correct position in renal artery, successfully performed renal nerve ablation procedure and has no related complications such as renal arterial perforation
Success rate of clinical treatment | 7 days after the procedure or at the time the patient is discharged from hospital
  based on succeed performance of renal interventional therapy procedure , there are no the procedure-related SAE, such as acute infection and renal dysfunction
All-cause death | 1 month, 3 months, 6 months, 9 months, 12 months, 24months, 36 months, 48 months and 60 months
Severe renal dysfunction | 6 months, 24months, 36 months, 48 months and 60 months
  eGFR<15mL/min/m2 or renal function replacement therapy needed
Rate of renal artery stenosis assessed by CT angiography | 6 months, 24months, 36 months, 48 months and 60 months
  (stenosis > 70% )
AEs, SAEs, and severe cardio-cerebrovascular events | 1 month, 3 months, 6 months, 9 months, 12months, 24months, 36 months, 48 months and 60 months
Reduction in 24-hour ABPM in systolic and diastolic arterial blood pressure | 24, 36, 48, 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Yong HUO, MD, Principal Investigator — Peking University First Hospital
Locations (15):
- China (15):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The Second Afflicted Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Norman Bethune International Peace Hospital, Shijiazhuang, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Shanghai Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Taiyuan Central Hospital, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin First Center Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided
Our decision on whether to share the individual participant data depends on the opinions of the regulatory authorities in China, but so far the regulatory agencies have no clear instructions yet, thus we cannot make a decision at present.

REFERENCES:
- [Derived] Wang J, Yin Y, Lu C, Lu Z, Hu J, Wang Y, Ge J, Jiang H, Yao C, Yan X, Ma W, Qi X, Dang Y, Chen S, Zhu J, Wang D, Ding C, Wang W, Liu J, Wang Y, Li H, Pan Z, Cui K, Li C, Liang X, Chen W, Sobotka PA, Zhang J, Esler M, Sun N, Chen M, Huo Y. Efficacy and safety of sympathetic mapping and ablation of renal nerves for the treatment of hypertension (SMART): 6-month follow-up of a randomised, controlled trial. EClinicalMedicine. 2024 May 7;72:102626. doi: 10.1016/j.eclinm.2024.102626. eCollection 2024 Jun. PMID 38756107
- [Derived] Wang J, Sun N, Ge J, Jiang H, Yin Y, Chen M, Wang Y, Yao C, Yan X, Sobotka PA, Huo Y. Rationale and Design of Sympathetic Mapping/Ablation of Renal Nerves Trial (SMART) for the Treatment of Hypertension: a Prospective, Multicenter, Single-Blind, Randomized and Sham Procedure-Controlled Study. J Cardiovasc Transl Res. 2023 Apr;16(2):358-370. doi: 10.1007/s12265-022-10307-z. Epub 2022 Aug 30. PMID 36042146
- [Derived] Wang Y, Wang JW, Wang Y, Yang B, Yinghua Du A, Kong Z, Chen M, Wang J. Monitoring Antihypertensive Medication Adherence by Liquid Chromatography-Tandem Mass Spectrometry: Method Establishment and Clinical Application. J Cardiovasc Pharmacol. 2021 Oct 1;78(4):581-596. doi: 10.1097/FJC.0000000000001105. PMID 34269698